CLINICAL TRIAL: NCT02827669
Title: One Drop Experts Program for Type 2 Diabetes Self-Management: Impact on A1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: One Drop (Unknown)
Responsible Party: Principal Investigator, Jessie Juusola, Sr. Director, Health Outcomes Research, Evidation Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EH-001
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- One Drop Experts Program (Experimental): Participants will be able to use the One Drop mobile app and One Drop Experts program on their smartphones. The One Drop mobile app is a diabetes management platform that allows users to track and log their blood glucose levels, medications, food, and activities. One Drop Experts is a diabetes education and coaching program delivered entirely through the One Drop mobile application.
  Interventions: Behavioral: One Drop Experts Program
- One Drop Experts Program + Apple Watch (Experimental): An Apple Watch will be provided to study participants in this arm. In addition to using the One Drop mobile app and One Drop Experts program on their smartphones, participants will also be able to engage with the app and program on their Apple Watch.
  Interventions: Behavioral: One Drop Experts Program + Apple Watch

INTERVENTIONS:
Behavioral: One Drop Experts Program
  Arms: One Drop Experts Program
Behavioral: One Drop Experts Program + Apple Watch
  Arms: One Drop Experts Program + Apple Watch

SUMMARY:
The One Drop Experts Program for Type 2 Diabetes Self-Management Impact on A1c trial is a 12-week long, prospective, intent-to-treat study that aims to evaluate the impact of the One Drop app and Experts program on HbA1c levels for individuals with uncontrolled Type 2 diabetes. A secondary objective will be to evaluate participants who utilize an Apple Watch in combination with the One Drop app and Experts program, and assess whether this group is more engaged or experiences a different impact as compared to participants who utilized the One Drop app and Experts program only.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Type 2 diabetes diagnosis
* Has not changed treatment regimen in the last 3 months
* HbA1c levels ≥ 7.5% by self-report and verified by lab test
* Motivated to use a daily diabetes self-management coaching program to improve diabetes control
* Owns and uses an iPhone with a compatible iOS operating system and has successfully downloaded and used a smartphone application previously

Exclusion Criteria:

* Current use of a smartphone application to manage their diabetes
* Currently participating in a diabetes self-management education or coaching program
* Currently pregnant
* Does not understand English
* History of serious mental illness or dementia
* Has severe diabetic complications such as severe diabetic retinopathy, chronic kidney disease (stages 4-5), severe diabetic neuropathy, diabetic foot ulcer or infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States